CLINICAL TRIAL: NCT06963541
Title: Comparison of IL-40 and IL-41 Levels in Patients With Sepsis and Septic Shock to Healthy Individuals
Brief Title: IL-40 and IL-41 Levels in Sepsis, Septic Shock, and Healthy Individuals
Status: Not yet recruiting | Type: Observational
Sponsor: Melahat Yalcin Solak (Other)
Responsible Party: Sponsor-Investigator, Melahat Yalcin Solak, lecturer doctor, Harran University
Organization: Harran University (Other)
Other Study IDs: HRÜ.27.01.25
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Sepsis; Septic Shock; Inflammation; Biomarkers
Keywords: IL-40; IL-41; Cytokines; Critical Illness; Septic Shock; Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic; Inflammation; Critical Illness | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis or Septic Shock Group: This cohort will include patients diagnosed with sepsis or septic shock based on the Sepsis-3 criteria. A one-time blood sample will be collected from each participant to analyze serum IL-40 and IL-41 levels. No intervention will be administered.
  Interventions: Other: No intervention; Observational study
- Healthy Control Group: Healthy volunteers with no history of chronic disease or recent infection. A single blood sample will be collected to measure baseline IL-40 and IL-41 levels.
  Interventions: Other: No intervention; Observational study

INTERVENTIONS:
Other: No intervention; Observational study — No interventions are associated with either group. This is an observational study without experimental procedures.

SUMMARY:
This study aims to investigate the blood levels of two recently identified immune-related proteins, Interleukin-40 (IL-40) and Interleukin-41 (IL-41), in patients with sepsis and its more severe form, septic shock. Sepsis is a serious condition caused by an abnormal immune response to infection, which can lead to organ dysfunction. Septic shock represents an advanced stage of sepsis, characterized by significantly higher mortality risk.

IL-40 and IL-41 are newly discovered molecules that are thought to play important roles in the immune system. In this study, the blood concentrations of IL-40 and IL-41 in patients diagnosed with sepsis or septic shock will be measured and compared with those in healthy individuals. The findings may contribute to understanding whether these proteins can be used as biomarkers in the diagnosis or monitoring of treatment in sepsis-related conditions.

DETAILED DESCRIPTION:
Sepsis is defined as a life-threatening organ dysfunction caused by a dysregulated host response to infection and is evaluated by an increase of two or more points in the Sequential Organ Failure Assessment (SOFA) score. Septic shock is characterized by hypotension that persists despite adequate fluid resuscitation (mean arterial pressure ≤65 mmHg) and a serum lactate level greater than 2 mmol/L. Septic shock represents a more severe clinical condition, with mortality rates reaching up to 60%.

Interleukin-40 (IL-40) is a recently discovered pro-inflammatory cytokine encoded by the chromosome 17 open reading frame 99 (C17orf99) gene. It is primarily produced by bone marrow, fetal liver, and activated peripheral B cells. IL-40 plays an essential role in immunoglobulin A production, humoral immune regulation, and B cell development. It has also been implicated in the pathogenesis of inflammatory diseases such as rheumatoid arthritis.

Interleukin-41 (IL-41), also known as meteorin-like protein (Metrnl), was identified in 2004 and is encoded by the meteorin-like (METRNL) gene located on chromosome 17q25.3. IL-41 is an anti-inflammatory cytokine expressed in tissues such as the intestines, skin, respiratory tract, and central nervous system. It is secreted primarily by alternatively activated macrophages and M2-like macrophages and has roles in both innate and adaptive immune responses.

The roles of IL-40 and IL-41 in sepsis and septic shock have not yet been fully elucidated. Understanding the involvement of these novel cytokines in inflammatory processes may provide new insights into the diagnosis and treatment of critical conditions such as sepsis and septic shock. The aim of this study is to compare IL-40 and IL-41 levels in patients diagnosed with sepsis or septic shock to those of healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patient Group:

Clinical diagnosis of sepsis or septic shock, based on validated diagnostic criteria (e.g., Sepsis-3)

Age 18 years or older

Ability and willingness to provide a blood sample prior to initiation of antibiotic treatment

Healthy Control Group:

Determined to be in good general health based on physical examination and medical history

Age 18 years or older

Willingness to provide written informed consent

Exclusion Criteria:

* Patient Group:

History of chronic inflammatory diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus)

Active cancer or current use of immunosuppressive therapy

Pregnant or breastfeeding

Presence of other serious conditions that may interfere with diagnosis or treatment (e.g., liver failure, chronic kidney disease)

Healthy Control Group:

Recent infection within the past month or use of antibiotics in the last 6 weeks

History of chronic inflammatory diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus)

Underwent surgery within the past 6 months

Conditions that may affect blood parameters, such as recent blood donation or intense physical activity

Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of two cohorts: (1) patients diagnosed with sepsis or septic shock based on Sepsis-3 criteria, and (2) healthy adult volunteers. Patients will be recruited from intensive care units and emergency departments, prior to the initiation of antibiotic therapy. Healthy controls will be selected based on clinical evaluation and medical history, confirming the absence of acute or chronic illness. All participants will be aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Serum IL-40 Levels Between Patients With Sepsis or Septic Shock and Healthy Controls | At time of enrollment (single time point)
  IL-40 concentration will be measured in serum samples from both groups using an ELISA-based method. The mean IL-40 levels will be compared between sepsis/septic shock patients and healthy individuals.
Comparison of Serum IL-41 Levels Between Patients With Sepsis or Septic Shock and Healthy Controls | At time of enrollment (single time point)
  IL-41 concentration will be measured in serum samples from both groups using an ELISA-based method. The mean IL-41 levels will be compared between sepsis/septic shock patients and healthy individuals.

SECONDARY OUTCOMES:
Correlation Between IL-40 and IL-41 Levels in All Participants | At time of enrollment (single time point)
  The study will assess the correlation between serum IL-40 and IL-41 levels among all participants, including both patient and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University Faculty of Medicine, Department of Anesthesiology and Reanimation, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical considerations, limited sample size, and absence of a formal data-sharing infrastructure.

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Cai S, Li X, Zhang C, Jiang Y, Liu Y, He Z, Ma S, Yao Y, Wong CK, Wu G, Gao X. Inhibition of Interleukin-40 prevents multi-organ damage during sepsis by blocking NETosis. Crit Care. 2025 Jan 16;29(1):29. doi: 10.1186/s13054-025-05257-2. PMID 39819454